CLINICAL TRIAL: NCT03292510
Title: Getting Older Adults OUTdoors (GO-OUT): A Randomized Controlled Trial of a Theory-based, Task-oriented, Outdoor Walking Program for Older Adults With Difficulty Walking Outdoors
Brief Title: Getting Older Adults OUTdoors (GO-OUT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University of Manitoba (Other); University of Alberta (Other); McGill University (Other)
Responsible Party: Principal Investigator, Dr. Nancy Salbach, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G-16-00013978
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Older Adults With Decreased Outdoor Walking Ability

STUDY DESIGN:
Intervention Model Description: Experimental: GO-OUT program An outdoor walking workshop with stations to learn various outdoor walking skills and information, followed by a supervised, group based outdoor walking program, twice a week for 60 minutes, for 10 weeks.
  Intervention: Other: GO-OUT program Active Comparator: Task-oriented outdoor walking workshop An outdoor walking workshop with stations to learn various outdoor walking skills and information.
  Intervention: Other: Task-oriented outdoor walking workshop
Who Masked: Outcomes Assessor
Masking Description: A 2-group mixed methods stratified randomized controlled trial following CONSORT criteria is proposed. Group allocation will be concealed and outcome evaluation blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GO-OUT Group (Experimental): Participants attend 1-day walking workshop followed by a 3-month outdoor walking group intervention, twice weekly for 60-minutes. The same activities are completed during both sessions within the same week. Each session includes a 10-minute warm-up, a distance walk, practice of a specific outdoor walking skill, a distance walk, and a 10-minute cool down. The warm up and cool down include stretching, functional strengthening exercises and balance exercises taught during the workshop. The program incorporates the principles of task-specific training by emphasizing repetitive practice of progressively more difficult outdoor walking tasks. The outdoor walking program is conducted in one or more large park settings given the mental health benefits of exercising in a natural environment.
  Interventions: Other: GO-OUT Group
- Workshop Group (Active Comparator): The 1-day workshop will be 5 hours with breaks. Participants will complete a series of stations learning information, strategies and skills related to safely walking outdoors. Stations include: pedometer use; walking pole use; footwear; footcare; fall prevention; balance exercises; proper use of walking aids; correct posture; self-management of exercise intensity; goal setting; and walking safely outdoors. Participants will receive a workbook with Canadian Physical Activity Guidelines, benefits of outdoor walking, information for each workshop station and a pedometer. Participants will use the workbook as an information resource and to record their community ambulation goals, planning routes, and walking time. All participants will be encouraged to walk outside with a partner, for safety.
  Interventions: Other: Workshop Group

INTERVENTIONS:
Other: GO-OUT Group — Following a baseline assessment, eligible participants will be stratified by site, and randomly assigned to receive the 1-day educational workshop and 3-month outdoor mobility program (GO-OUT intervention). Follow-up evaluations will occur at 3, 5.5 and 12 months from baseline.
  Arms: GO-OUT Group
Other: Workshop Group — the 1-day workshop plus reminders. Follow-up evaluations will occur at 3, 5.5 and 12 months from baseline
  Arms: Workshop Group

SUMMARY:
Community walking is an issue that older adults with chronic conditions have described as important to participation in the community. Walking outside the home is a universally accessible form of physical activity that has multiple health benefits. Walking for 150 minutes per week can help reduce the risk of cardiovascular disease, hypertension, stroke, diabetes, osteoporosis, and depression, as well as falls. Practice walking across roads, slopes and curbs, while talking, and dealing with crowds and traffic, is safe and feasible and can improve confidence, balance and walking ability. Being physically active outdoors in nature appears to improve mental health more than being active indoors. Despite these health benefits, the majority of older Canadians do not walk outside on a regular basis. Barriers to walking outside include fear, physical disability due to chronic disease, the appropriateness of footwear and walking aids, and the physical environment, such as uneven pavement, weather and temperature. To date, the best strategy for getting people to walk outdoors regularly is unknown. The investigators propose to evaluate the effectiveness of a dynamic 1-day workshop, at which older adults who infrequently walk outdoors learn strategies to facilitate outdoor walking, such as appropriate use of footwear, ambulatory aids and equipment, goal setting, and practice skills related to increasing outdoor walking. The workshop will be compared to the workshop plus involvement in a walking group for 3 months. Outcomes include outdoor walking activity, total physical activity, walking ability, participation, and health-related quality of life. Each participant will have four evaluations: baseline, 3, 5.5 and 12 months later. The investigators will interview select participants at 6 and 12 months to ask them about their opinions of what worked and didn't work. Increasing outdoor walking is expected to improve health and well-being, and help people live independently in the community for longer.

DETAILED DESCRIPTION:
Background: Inability to walk outdoors restricts full participation in physical activity and community living for older adults that can reduce health-related quality of life (HRQL). Older adults report limited outdoor walking with only 8% achieving the Canadian recommendation for older adults of 150 minutes of moderate-to-vigorous (MV) intensity physical activity per week. Known barriers to walking outside include fear, physical disability due to chronic disease, the appropriateness of footwear and walking aids, the physical environment, weather and temperature. Group practice walking outdoors in locations with variable environmental challenges has the potential to improve physical ability, confidence, outdoor and overall physical activity and social participation. The extent to which it is safe and feasible to implement this intervention in people with varying degrees of physical ability, preferences for where to walk, neighbourhood walkability, and to measure outdoor walking activity, is unclear.

Objectives: In older adults with a limitation in outdoor community mobility:

1. To estimate the extent to which a 1-day educational workshop and 10-week outdoor mobility program (GO-OUT intervention) compared to the workshop and weekly reminders improves outdoor walking activity (primary outcome) and secondary outcomes of physical activity, lifespace mobility, participation, HRQL, balance, leg strength, walking self-efficacy, walking speed, walking distance/endurance, and mood over 12 months.
2. To explore participants' perceptions of intended and unintended consequences of the interventions, potent intervention components, mechanisms of effect, modifying influences of disability level, sex,neighborhood walkability, weather, car access, and study site, and recommendations for future program delivery models.

Approaches and Methods:Study Design: A 2-group mixed methods stratified randomized controlled trial following CONSORT criteria is proposed. Group allocation will be concealed and outcome evaluation blinded. The trial will be run at 4 sites (Edmonton, Winnipeg, Toronto, Montreal) to accrue a sufficient sample size, optimize the external validity of the results to urban centres variable in population size, weather conditions, and environmental barriers, and build capacity across 4 provinces to support potential implementation. Following a baseline assessment, eligible participants will be stratified by site, and randomly assigned to receive the 1-day educational workshop and 3-month outdoor mobility program (GO-OUT intervention) or the 1-day workshop plus weekly reminders. Follow-up evaluations will occur at 3, 5.5 and 12 months from baseline. A sub-sample of participants from the GO-OUT and workshop groups at each site will participate in face-to-face interviews at 6 and 12 months to explore their experiences. Interventions and assessments are designed to be implemented in 'good weather' months, to avoid the potential negative effect of season on the primary outcome of outdoor walking activity.

ELIGIBILITY:
Inclusion Criteria:

1. older adults defined as age 65 years or older;
2. living independently in the community;
3. ambulatory defined as self-reported ability to walk at least one block (~50 m) continuously on a flat surface with or without a walking aid and without supervision;
4. self-reported difficulty walking in the outdoor community environment (this could include physical impairments or decreased confidence);
5. willingness to sign a liability waiver (required at three sites) or send a letter to their physician (required at one site) regarding clearance to exercise;
6. mental competency defined by a score of at least 18 out of 22 on the Mini-Mental State Exam telephone version;
7. available for a scheduled workshop and at least 5 of 10 weeks of the outdoor walking program; and
8. ability to speak and understand English

Exclusion Criteria:

1. physically active defined as self-reported participation in physical activities, such as walking and playing golf, 150 min per week;
2. currently receiving rehabilitation treatment, such as physical or occupational therapy, for goals related to walking (self-report);
3. at high falls risk defined by meeting one or more of the following American Geriatric Society criteria: (A) ≥2 falls in the last 12 months or presents with an acute fall; (B) cardiac, respiratory, peripheral vascular or other health conditions that would prevent safe and full participation in the interventions (self-report); (C) postural hypotension defined as a drop in systolic BP of >20 mm Hg or a drop in diastolic BP of >10 mm Hg taken after lying supine for 5 min and after standing for 2 min; (D) resting HR <45 or >100 beats per minute; and (E) severe limitation in visual acuity defined as self-reported difficulty reading the newspaper while wearing regular reading glasses or bifocals, or self-reported inability to distinguish a person's facial features from across a room while wearing glasses.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in average number of minutes per week spent walking outdoors | baseline, 3, 5.5, 12 months
  The ActiGraph GT3X+ activity monitor (www.actigraphcorp.com/products/wgt3x-monitor/, ActiGraph, Pensacola, FL) and Qstarz BT-Q1000XT A-GPS Travel Recorder (http://www.qstarz.com/Products/GPS%20Products/BT-Q1000XT-F.htm) will be worn by each participant, clipped onto their waist band over the right hip during waking hours for 8 consecutive days at each evaluation timepoint (baseline, 3, 5.5, and 12 months).

SECONDARY OUTCOMES:
Change in the mean time per week spent walking outdoors on the Community Health Activities Model Program for Seniors (CHAMPS) Questionnaire | baseline, 3, 5.5, 12 months
  The Community Health Activities Model Program for Seniors (CHAMPS) questionnaire is a measure of participation, physical activity and outdoor walking. Participants self-report time spent performing various social, leisure, and physical activities in a typical week during the last 4 weeks. Total time spent per week in outdoor walking will be determined.
Change in the mean time per week spent in meaningful activity on the Community Health Activities Model Program for Seniors (CHAMPS) Questionnaire | baseline, 3, 5.5, 12 months
  The Community Health Activities Model Program for Seniors (CHAMPS) questionnaire is a measure of participation, physical activity and outdoor walking. Participants self-report time spent performing various social, leisure, and physical activities in a typical week during the last 4 weeks. Total time spent per week in any activity will be determined.
Change in the mean self-reported time per week spent in moderate- to vigorous-intensity physical activity on the Community Health Activities Model Program for Seniors (CHAMPS) Questionnaire | baseline, 3, 5.5, 12 months
  The Community Health Activities Model Program for Seniors (CHAMPS) questionnaire is a measure of participation, physical activity and outdoor walking. Participants self-report time spent performing various social, leisure, and physical activities in a typical week during the last 4 weeks. Total time spent per week in moderate- to vigorous-intensity aerobic physical activity is determined.
Change in the mean time per week spent in moderate- to vigorous-intensity physical activity directly measured using ActiGraph and GPS devices | baseline, 3, 5.5, 12 months
  The ActiGraph GT3X+ activity monitor (www.actigraphcorp.com/products/wgt3x-monitor/, ActiGraph, Pensacola, FL) and Qstarz BT-Q1000XT A-GPS Travel Recorder (http://www.qstarz.com/Products/GPS%20Products/BT-Q1000XT-F.htm) will be worn by each participant, clipped onto their waist band over the right hip during waking hours for 8 consecutive days at each evaluation timepoint (baseline, 3, 5.5, and 12 months).
Change in the mean score on the Life Space Assessment Questionnaire | baseline, 3, 5.5, 12 months
  The Life Space Assessment Questionnaire is a measure of life space mobility. Total scores can range from 0 (totally bed bound) to 120 (travels out of the city every day without assistance). The score indicates level, degree of independence and frequency of attainment of mobility in five living spaces in the past four weeks: rooms in the house, the area outside the house, places in the neighbourhood, places outside the neighbourhood but within the city, and places outside the city.
Change in the mean scores on the Patient Generated Index (PGI) | baseline, 3, 5.5, 12 months
  For the PGI, participants select five most important areas of their life that are affected by their health, then rates the degree to which each area is affected from 0 (worst level imaginable) to 10 (best level of function possible).
Change in the mean scores on the Research ANd Development-36 (RAND-36) | baseline, 3, 5.5, 12 months
  The RAND-36 is a 36-item self-report measure of 8 health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain and general health perceptions. Total scores range from 0 to 100, where higher scores represent the most optimal health state.
Change in the mean total score on the Mini Balance Evaluations Systems Test (Mini BESTest) | baseline, 3, 5.5, 12 months
  The Mini BESTest is a measure of balance. Total scores can range from 0 to 28 points.
Change in the mean number of sit-to-stands completed in 30 seconds in the 30-second Sit to Stand Test. | baseline, 3, 5.5, 12 months
  The 30-second Sit to Stand Test is a measure of lower extremity strength. The minimum score is 0.
Change in the mean score on the Ambulatory Self-Confidence Questionnaire | baseline, 3, 5.5, 12 months
  The Ambulatory Self-Confidence Questionnaire is a 22-item questionnaire to measure self-efficacy to walk at home and/or in the community. The total score is the mean of item-level scores and can range from 0 to 10.
Change in the mean walking speed on the 10m Walk Test, completed at a comfortable pace and a fast pace | baseline, 3, 5.5, 12 months
  The 10m Walk Test is a measure of the participant's walking speed at a comfortable and fast pace. The participant uses his/her usual assistive device(s) and corrective eyewear.
Change in the mean distance (in metres) walked on the 6-Minute Walk Test | baseline, 3, 5.5, 12 months
  The 6-Minute Walk Test is a measure of walking endurance. Participants walk for 6 minutes unassisted using his/her usual mobility device. The distance walked in metres in 6 minutes is recorded.
Change in resting heart rate | baseline, 3, 5.5, 12 months
  Heart rate (HR) is taken at rest after sitting for at least 5 minutes with back supported and feet flat on the floor. HR is taken through manual palpation of the radial artery for 1 minute. Resting HR is part of the screening for participants prior to administering the 6-Minute Walk Test.
Change in resting blood pressure | baseline, 3, 5.5, 12 months
  Blood pressure (BP) is taken at rest after sitting for at least 5 minutes with back supported and feet flat on the floor. BP is taken using a manual or automated documented. Resting BP is part of the screening for participants prior to administering the 6-Minute Walk Test.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Salbach, PhD, Principal Investigator — Associate Professor
Locations (1):
- Knowledge to Action Lab, Department of Physical Therapy, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kokorelias KM, Ripat J, Barclay R, Jones CA, Mayo NE, Grant T, Scodras S, Alsbury-Nealy K, Ryder-Burbidge C, Salbach NM. A park-based group mobility program for older adults with difficulty walking outdoors: a qualitative process evaluation of the Getting Older Adults Outdoors (GO-OUT) randomized controlled trial. BMC Geriatr. 2025 Jan 8;25(1):16. doi: 10.1186/s12877-024-05611-z. PMID 39780066
- [Derived] Salbach NM, Mayo NE, Webber SC, Jones CA, Lix LM, Ripat J, Grant T, van Ineveld C, Chilibeck PD, Romanescu RG, Scott S, Barclay R. Short-term effects of a park-based group mobility program on increasing outdoor walking in older adults with difficulty walking outdoors: the Getting Older Adults Outdoors (GO-OUT) randomized controlled trial. BMC Geriatr. 2024 Sep 6;24(1):740. doi: 10.1186/s12877-024-05331-4. PMID 39243012
- [Derived] Barclay R, Webber SC, Hahn F, Jones CA, Mayo NE, Sivakumaran S, Liu Y, Chilibeck PD, Salbach NM. A park-based group mobility program for older adults with difficulty walking outdoors: a quantitative process evaluation of the Getting Older Adults Outdoors (GO-OUT) randomized controlled trial. BMC Geriatr. 2023 Dec 11;23(1):833. doi: 10.1186/s12877-023-04524-7. PMID 38082248
- [Derived] Salbach NM, Barclay R, Webber SC, Jones CA, Mayo NE, Lix LM, Ripat J, Grant T, van Ineveld C, Chilibeck PD. A theory-based, task-oriented, outdoor walking programme for older adults with difficulty walking outdoors: protocol for the Getting Older Adults Outdoors (GO-OUT) randomised controlled trial. BMJ Open. 2019 Apr 20;9(4):e029393. doi: 10.1136/bmjopen-2019-029393. PMID 31005945